CLINICAL TRIAL: NCT01599858
Title: YF476: Effects of Repeated Dosing at 2 Dose Levels on 24-hour Ambulatory Gastric pH Compared With Placebo and Omeprazole in Healthy Volunteers
Brief Title: Effect of Repeated Doses of YF476, Omeprazole and Placebo on Stomach Acidity in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 96-018
Record Dates: First submitted 2012-05-10; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Reflux Oesophagitis
Keywords: YF476; gastrin receptor antagonist; gastric pH; healthy subjects; omeprazole
MeSH Terms: conditions — Esophagitis, Peptic | interventions — YF 476; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YF476 — There were 4 treatments as follows: YF476 25mg twice daily, YF476 100mg twice daily, placebo and omeprazole 20mg once daily. Each treatment was taken by mouth for 7 days. Each subject took 1 of the 4 treatments.
Drug: Omeprazole — There were 4 treatments as follows: YF476 25mg twice daily, YF476 100mg twice daily, placebo and omeprazole 20mg once daily. Each treatment was taken by mouth for 7 days. Each subject took 1 of the 4 treatments.

SUMMARY:
The objectives of this study were:

To compare repeated doses of YF476 at 2 dose levels, placebo and omeprazole with respect to their effect on basal- and food- stimulated gastric pH in healthy volunteers.

To compare repeated doses of YF476 at 2 dose levels, placebo and omeprazole with respect to their effect on basal and meal stimulated pH.

To assess the safety, tolerability and pharmacokinetics of repeated doses of YF476 in healthy volunteers.

DETAILED DESCRIPTION:
YF476 is clearly a potent and selective gastrin/CCK-B antagonist and should inhibit basal and meal-stimulated gastric acid secretion, enhance gastric emptying of a liquid meal and increase lower oesphageal sphincter pressure in man. Therefore YF476 might benefit patients with reflux oesophagitis.

YF476 has been well tolerated in healthy volunteers at single doses up to 100mg and remarkably well tolerated at repeat doses in animals up to 350 times the maximum dose planned for the proposed study. A range of doses of YF476 (25 and 100mg twice daily) will be administered to steady state. 24-hour ambulatory gastric pH will be monitored via an intragastric pH electrode to assess the effect of YF476 on basal and meal stimulated gastric pH. Although there is variability between subjects with respect to the effects of food and drug treatment on gastric pH, the methodology for measurement of ambulatory gastric pH is robust.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-45 years.
* No clinically relevant abnormal findings in the clinical history or physical examination at the screening assessment which could interfere with the objectives of the study or make the subject's participation hazardous.
* No clinically relevant abnormal laboratory values at the screening evaluation (Attachment 2).
* A normal ECG at the screening examination.
* A body mass index (Quetelet index) in the range 19-30:

Body Mass Index = weight [kg]_ height [m]2

* Normal blood pressure and heart rate at the screening examination, i.e. BP 90-150mmHg systolic, 40-95mmHg diastolic; heart rate 40-100 beats/min in seated position.
* Subjects must be of sufficient intelligence to understand the nature of the study and any hazards of their participation in it. They must be able to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Subjects must give their written consent to participate after reading the Information-for-Volunteers Leaflet and Consent Form, and after having the opportunity to discuss the study with the Investigator or his deputy.

Exclusion Criteria:

* Females who are pregnant or lactating, or who are sexually active and are not using a reliable method of contraception.
* Clinically relevant abnormal history or physical findings at the screening assessment, which could interfere with the objectives of the study or the safety of the subject's participation.
* Clinically relevant abnormalities of laboratory values or ECG at screening evaluation.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate subject's participation in the study or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease or history of any psychotic mental illness.
* Participation in other clinical studies of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 40 units of alcohol weekly.
* Loss of more than 400mL blood during the 3 months before the study, e.g. as a blood donor.
* Use of prescription medication during 30 days before the study.
* Use of an over-the-counter medicine during 7 days before the study
* Blood pressure or heart rate outside those values specified under inclusion criterion (f).
* Possibility that the subject will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing at study entry.
* Positive test for hepatitis B or C or HIV 1 & 2.
* High risk of hepatitis or HIV infection.
* History of severe allergic disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 1996-08; Primary Completion 1996-10 (Actual); Study Completion 1996-10 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic measurements: continuous 24h ambulatory gastric pH and 24 h plasma gastrin | 6 weeks
  Recording started 0.5 h before the morning dose on Study Day 7 for measurement of gastric pH; meals taken at 4, 9, 13 & 22 h after the morning dose. Frequent blood samples for measurement of plasma gastrin.
Assessment of safety and tolerability | 6 weeks
  Physical examination, ECG and safety tests of blood/urine at screening, after the last dose and at follow up.
Pharmacokinetic analysis of plasma YF476 concentrations | 6 weeks
  Blood samples (8 mL) for assay of YF476 taken before each morning dose on Study Days 1-6 and at 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 12.25, 12.5, 12.75, 13, 14.5, 15, 16, 17, 18, 20, 22 and 24h on Study Day 7 (where 0h is the time of the morning dose and 12h is the time of the evening dose)for calculation of Cmax, Tmax, AUC 0-24 h, T1/2.
Number of adverse events | 6 weeks
  Adverse events throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Study Director — Trio Medicines Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom